CLINICAL TRIAL: NCT00392327
Title: Efficacy of Carboplatin Administered Concomitantly With Radiation and Isotretinoin as a Pro-Apoptotic Agent in Other Than Average Risk Medulloblastoma/PNET Patients
Brief Title: Chemotherapy and Radiation Therapy in Treating Young Patients With Newly Diagnosed, Previously Untreated, High-Risk Medulloblastoma/PNET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0332; NCI-2009-00336 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07-271; CDR0000511991; COG-ACNS0332; ACNS0332 (Other: Children's Oncology Group); ACNS0332 (Other: CTEP); R01CA114567 (NIH); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Anaplastic Medulloblastoma; Medulloblastoma
MeSH Terms: conditions — Medulloblastoma | interventions — Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Isotretinoin; Spinal Puncture; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (chemoradiotherapy) (Active Comparator): CHEMORADIOTHERAPY: Patients undergo radiation therapy QD five days a week for 6 weeks. Patients also receive vincristine sulfate IV over 1 minute once weekly for 6 weeks. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.
  MAINTENANCE THERAPY: Patients receive cisplatin IV over 6 hours on day 1, vincristine sulfate IV over 1 minute on days 1 and 8, and cyclophosphamide IV over 1 hour on days 2 and 3. Patients also receive filgrastim SC or IV beginning on day 4 and continuing until blood counts recover (at least 10 days).
  Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.
  Patients also undergo blood sample collection, lumbar puncture and MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Drug: Cyclophosphamide; Biological: Filgrastim; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Arm B (chemoradiotherapy) (Experimental): CHEMORADIOTHERAPY: Patients receive vincristine sulfate and undergo radiation therapy as in Arm A. Patients also receive carboplatin IV over 15 minutes on each day of radiation therapy. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.
  MAINTENANCE THERAPY: Patients receive maintenance therapy as in Arm A.
  Patients also undergo blood sample collection, lumbar puncture and MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Biological: Filgrastim; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Arm C (chemoradiotherapy, isotretinoin-CLOSED TO ACCRUAL) (Experimental): CHEMORADIOTHERAPY: Patients undergo chemoradiotherapy as in Arm A. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.
  MAINTENANCE THERAPY: Patients receive isotretinoin PO BID on day 1 and days 16-28 and cisplatin, vincristine sulfate, cyclophosphamide, and filgrastim as in Arm A maintenance therapy. Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive isotretinoin PO BID on days 15-28 every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Cyclophosphamide; Biological: Filgrastim; Drug: Isotretinoin; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate
- Arm D (chemoradiotherapy, isotretinoin-CLOSED TO ACCRUAL) (Experimental): CHEMORADIOTHERAPY: Patients undergo chemoradiotherapy as in Arm B. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.
  MAINTENANCE THERAPY: Patients receive maintenance therapy as in Arm C. Patients then proceed to continuation therapy.
  CONTINUATION THERAPY: Patients receive continuation therapy as in Arm C.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Cyclophosphamide; Biological: Filgrastim; Drug: Isotretinoin; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Drug: Vincristine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm A (chemoradiotherapy); Arm B (chemoradiotherapy)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm B (chemoradiotherapy); Arm D (chemoradiotherapy, isotretinoin-CLOSED TO ACCRUAL)
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Biological: Filgrastim — Given IV or SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Drug: Isotretinoin — Given PO
  Other Names: 13-cis retinoic acid; 13-cis-Retinoate; 13-cis-Retinoic Acid; 13-cis-Vitamin A Acid; 13-cRA; Absorica; Accure; Accutane; Amnesteem; cis-Retinoic Acid; Cistane; Claravis; Isotretinoinum; Isotrex; Isotrexin; Myorisan; Neovitamin A; Neovitamin A Acid; Oratane; Retinoicacid-13-cis; Ro 4-3780; Ro-4-3780; Roaccutan; Roaccutane; Roacutan; Sotret; ZENATANE
  Arms: Arm C (chemoradiotherapy, isotretinoin-CLOSED TO ACCRUAL); Arm D (chemoradiotherapy, isotretinoin-CLOSED TO ACCRUAL)
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
  Arms: Arm A (chemoradiotherapy); Arm B (chemoradiotherapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Arm A (chemoradiotherapy); Arm B (chemoradiotherapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies different chemotherapy and radiation therapy regimens to compare how well they work in treating young patients with newly diagnosed, previously untreated, high-risk medulloblastoma. Chemotherapy drugs, such as vincristine sulfate, cisplatin, cyclophosphamide, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Radiation therapy uses high-energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Carboplatin may make tumor cells more sensitive to radiation therapy. It is not yet known which chemotherapy and radiation therapy regimen is more effective in treating brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether carboplatin radiosensitization increases long term event-free survival for high risk medulloblastoma/primitive neuroectodermal tumor (PNET) patients.

II. To determine whether isotretinoin increases long term event-free survival for high risk medulloblastoma/PNET patients.

CORRELATIVE SCIENCE OBJECTIVES:

I. To compare residual disease response to radiation alone versus radiation plus carboplatin.

II. To identify molecular prognostic indicators suitable for patient stratification in future trials.

III. To evaluate the health-related quality of life (HRQOL) during phases of active treatment specific to treatment modalities.

IV. To describe the neuropsychological functioning of the study population and to evaluate the relationship between neuropsychological status and health related quality of life.

OUTLINE: Patients are randomized to Arm A or Arm B (Arms C and D closed to accrual as of Amendment 3 1/27/15).

ARM A (standard chemoradiotherapy and standard maintenance therapy):

CHEMORADIOTHERAPY: Patients undergo radiation therapy once daily (QD) five days a week for 6 weeks. Patients also receive vincristine sulfate intravenously (IV) over 1 minute once weekly for 6 weeks. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive cisplatin IV over 6 hours on day 1, vincristine sulfate IV over 1 minute on days 1 and 8, and cyclophosphamide IV over 1 hour on days 2 and 3. Patients also receive filgrastim subcutaneously (SC) or IV beginning on day 4 and continuing until blood counts recover (at least 10 days). Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients also undergo blood sample collection, lumbar puncture and magnetic resonance imaging (MRI) throughout the study.

ARM B (standard chemoradiotherapy plus carboplatin and standard maintenance therapy):

CHEMORADIOTHERAPY: Patients receive vincristine sulfate and undergo radiation therapy as in Arm I. Patients also receive carboplatin IV over 15 minutes on each day of radiation therapy. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive maintenance therapy as in Arm I.

Patients also undergo blood sample collection, lumbar puncture and MRI throughout the study.

ARM C (standard chemoradiotherapy, standard maintenance therapy plus isotretinoin, and continuation therapy with isotretinoin - CLOSED TO ACCRUAL 1/27/15):

CHEMORADIOTHERAPY: Patients undergo chemoradiotherapy as in Arm I. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive isotretinoin orally (PO) twice daily (BID) on day 1 and days 16-28 and cisplatin, vincristine sulfate, cyclophosphamide, and filgrastim as in Arm I maintenance therapy. Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to continuation therapy.

CONTINUATION THERAPY: Patients receive isotretinoin PO BID on days 15-28 every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM D (standard chemoradiotherapy plus carboplatin, standard maintenance therapy plus isotretinoin, and continuation therapy with isotretinoin - CLOSED TO ACCRUAL 1/27/15):

CHEMORADIOTHERAPY: Patients undergo chemoradiotherapy as in Arm II. Six weeks after completion of chemoradiotherapy, patients proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive maintenance therapy as in Arm III. Patients then proceed to continuation therapy.

CONTINUATION THERAPY: Patients receive continuation therapy as in Arm III.

After completion of study treatment, patients are followed up periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 3 and less than 22 years at the time of diagnosis
* Newly diagnosed, previously untreated: (1) M0 medulloblastoma with > 1.5 cm^2 residual; (2) M+ medulloblastoma; patients with diffusely anaplastic medulloblastoma are eligible regardless of M-stage or residual tumor

  * As of amendment # 2, enrollment of patients with supratentorial PNET has been discontinued
  * All patients with M4 disease are not eligible
* A pre-operative magnetic resonance imaging (MRI) scan of the brain with and without contrast is required; NOTE: computed tomography (CT) scans are NOT sufficient for study eligibility since radiation therapy planning and response will be based on MRI scans only

  * Post-operative head MRI scan with and without contrast (preferably within 72 hours post-surgery); for patients who undergo stereotactic biopsy only, either a pre or post-operative MRI is sufficient; for patients with M2 and M3 disease, a post-op MRI is strongly encouraged, but not mandatory
  * Spinal MRI imaging with and without gadolinium is required within 10 days of surgery if done pre-operatively or within 28 days of surgery if done post-operatively; for posterior fossa tumors, pre-operative MRI scans are preferred because surgically-induced inflammation/blood can be difficult to distinguish from tumor
* Lumbar cerebrospinal fluid (CSF) cytology examination must be obtained pre-operatively or within 31 days following surgery; the optimal time for obtaining CSF is prior to surgery or 1-3 weeks following surgery; ventricular CSF (either pre- or post-op) may be used only if a post-operative spinal tap is contraindicated; if a spinal tap is contraindicated and there is no ventricular CSF available, then CSF cytology can be waived for patients with supratentorial tumors or if there is documentation of spinal subarachnoid metastases (M3); patients who are categorized as M1 must have either an intra-operative positive CSF (via lumbar puncture at the end of the procedure) or a positive lumbar CSF obtained > 7 days post-operatively (to rule out surgically induced false positives)
* Patients must have a Karnofsky performance level of >= 30 for patients > 16 years of age or a Lansky performance scale of >= 30 for patients =< 16 years of age and life expectancy > 8 weeks
* No previous chemotherapy or radiation therapy
* Corticosteroids should not be used during chemotherapy administration as an antiemetic because of their effect on the blood-brain barrier
* Clinically significant drug interactions have been reported when using vincristine with strong CYP450 3A4 inhibitors and inducers. Selected strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (cytochrome P450 3A4) include azole antifungals, such as fluconazole, voriconazole, itraconazole, ketoconazole, and strong inducers include drugs such as rifampin, phenytoin, phenobarbitol, carbamazepine, and St. John's wort; the use of these drugs should be avoided with vincristine (vincristine sulfate)
* The clinical outcome and significance of CYP450 interactions with cyclophosphamide are less clear. CYP450 3A4 stimulators or inhibitors should be avoided or used with great caution; aprepitant also interacts with CYP3A4 and should be used with caution with etoposide or vincristine chemotherapy
* Cisplatin should be used with caution with nephrotoxic drug; aminoglycoside should be avoided or used with caution during or shortly after cisplatin administration and concomitant use with amphotericin B should probably also be avoided; patients receiving cisplatin and other potentially ototoxic drugs such as aminoglycoside or loop diuretics concomitantly should be closely monitored for signs of ototoxicity

  * In patients receiving cisplatin and phenytoin or fosphenytoin, serum concentrations of phenytoin may decrease. Carbamazepine concentration may also decrease with concomitant use. Plasma levels of anticonvulsant agents should be monitored and doses adjusted during therapy with cisplatin
* No other experimental therapy is permitted while on study
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Total bilirubin < 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age; for patients on anti-seizure medications, SGOT (AST) or SGPT (ALT) must be < 5 x ULN
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets >= 100,000/uL (untransfused)
* Hemoglobin >= 8 g/dl (may be transfused)
* There is information indicating a risk of fetal or teratogenic toxicity with this treatment. Female patients who are post-menarchal must have a negative pregnancy test; lactating female patients must agree not to breast-feed while on this trial; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 3 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 379 (Actual)
Dates: Start 2007-05-23 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2028-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Leary, Principal Investigator — Children's Oncology Group
Locations (185):
- United States (170):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Dutch Childhood Oncology Group, Utrecht, Netherlands
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Hwang EI, Kool M, Burger PC, Capper D, Chavez L, Brabetz S, Williams-Hughes C, Billups C, Heier L, Jaju A, Michalski J, Li Y, Leary S, Zhou T, von Deimling A, Jones DTW, Fouladi M, Pollack IF, Gajjar A, Packer RJ, Pfister SM, Olson JM. Extensive Molecular and Clinical Heterogeneity in Patients With Histologically Diagnosed CNS-PNET Treated as a Single Entity: A Report From the Children's Oncology Group Randomized ACNS0332 Trial. J Clin Oncol. 2018 Oct 17;36(34):JCO2017764720. doi: 10.1200/JCO.2017.76.4720. Online ahead of print. PMID 30332335
- [Derived] Leary SES, Packer RJ, Li Y, Billups CA, Smith KS, Jaju A, Heier L, Burger P, Walsh K, Han Y, Embry L, Hadley J, Kumar R, Michalski J, Hwang E, Gajjar A, Pollack IF, Fouladi M, Northcott PA, Olson JM. Efficacy of Carboplatin and Isotretinoin in Children With High-risk Medulloblastoma: A Randomized Clinical Trial From the Children's Oncology Group. JAMA Oncol. 2021 Sep 1;7(9):1313-1321. doi: 10.1001/jamaoncol.2021.2224. PMID 34292305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (Pts) 3-21 yrs were recruited at COG institutions.The first pt was enrolled 5/23/2007, and the last pt was enrolled 4/9/2018.The study was initially open to medulloblastoma and supratentorial primitive neuroectodermal tumor (SPNET) pts, but closed for SPNET pts as of amendment #2.All pts were off treatment at the time of results reporting.
Pre-assignment Details: Participants received standard therapy consisting of surgery, radiation and chemotherapy. A subset of patients was randomly assigned to receive carboplatin. A second randomization was used to randomly assign patients to receive isotretinoin. Of note, the isotretinoin randomization was stopped early due to futility.
Groups:
- Regimen A (Medulloblastoma Patients): Medulloblastoma patients who received regimen A (no carboplatin / no isotretinoin)
- Regimen B (Medulloblastoma Patients): Medulloblastoma patients who received regimen B (carboplatin / no isotretinoin)
- Regimen C (Medulloblastoma Patients): Medulloblastoma patients who received regimen C (no carboplatin / isotretinoin)
- Regimen D (Medulloblastoma Patients): Medulloblastoma patients who received regimen D (carboplatin / isotretinoin)
- Regimen A (SPNET Patients): SPNET patients who received regimen A (no carboplatin / no isotretinoin)
- Regimen B (SPNET Patients): SPNET patients who received regimen B (carboplatin / no isotretinoin)
- Regimen C (SPNET Patients): SPNET patients who received regimen C (no carboplatin / isotretinoin)
- Regimen D (SPNET Patients): SPNET patients who received regimen D (carboplatin / isotretinoin)
Period: Overall Study
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients) | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Started | 87 | 93 | 56 | 58 | 23 | 19 | 21 | 22
Completed | 72 | 74 | 36 | 42 | 20 | 14 | 12 | 11
Not Completed | 15 | 19 | 20 | 16 | 3 | 5 | 9 | 11
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 8 | 9 | 6 | 3 | 3 | 3 | 3
Not completed — Physician Decision | 3 | 5 | 2 | 2 | 0 | 1 | 5 | 3
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 4 | 6 | 0 | 1 | 1 | 5
Not completed — Ineligible | 0 | 4 | 3 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible patients were included in the baseline characteristics results. For example, of the 93 Regimen B medulloblastoma patients, 4 were ineligible (see patient flow) and excluded from baseline measures reporting leaving 89 eligible regimen B medulloblastoma patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients) | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients) | Total
Number analyzed (Participants) | 87 | 89 | 53 | 56 | 23 | 19 | 21 | 22 | 370
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 88 | 51 | 55 | 23 | 19 | 21 | 22 | 365
  Between 18 and 65 years | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8.2 [3.5 to 19.2] | 8.8 [3.5 to 21.2] | 9.1 [3.3 to 20.1] | 9 [3.4 to 19.9] | 10.7 [3.1 to 18.1] | 9.4 [3.5 to 16.9] | 8.9 [3.1 to 17.9] | 10.3 [3.0 to 17.6] | 8.8 [3.0 to 21.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 15 | 21 | 13 | 10 | 12 | 12 | 134
  Male | 65 | 60 | 38 | 35 | 10 | 9 | 9 | 10 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 10 | 13 | 3 | 4 | 2 | 2 | 53
  Not Hispanic or Latino | 75 | 79 | 41 | 42 | 20 | 15 | 18 | 19 | 309
  Unknown or Not Reported | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
  Asian | 1 | 4 | 3 | 1 | 0 | 2 | 3 | 0 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 7 | 5 | 0 | 9 | 2 | 3 | 8 | 46
  White | 63 | 69 | 38 | 49 | 13 | 13 | 10 | 12 | 267
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 10 | 8 | 6 | 6 | 1 | 2 | 4 | 2 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Probability of Event-free Survival (EFS) for Patients With Medulloblastoma
Description: The Kaplan-Meier method will be used to estimate 5-year EFS, defined as the time from study enrollment to disease progression or recurrence, second malignant neoplasm, or death from any cause, or to date of last contact. Estimates are reported with 95% confidence intervals. Data below represents all molecular subgroups combined.
Time Frame: Up to 5 years
Population: Eligible medulloblastoma patients are included.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients)
Number analyzed (Participants) | 87 | 89 | 53 | 56
Percent Probability | 57.5 [43.6 to 71.4] | 65.3 [52.0 to 78.6] | 60.3 [47.0 to 73.6] | 70.9 [57.8 to 84.0]

2. Primary Outcome: Percent Probability of Event-free Survival (EFS) for Patients With Supratentorial Primitive Neuroectodermal Tumor (SPNET)
Description: The Kaplan-Meier method will be used to estimate 5-year EFS, defined as the time from study enrollment to disease progression or recurrence, second malignant neoplasm, or death from any cause, or to date of last contact. Estimates are reported with 95% confidence intervals.
Time Frame: Up to 5 years
Population: Eligible SPNET patients are included.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 23 | 19 | 21 | 22
Percent Probability | 52.2 [32.6 to 71.8] | 52.6 [31.2 to 74.0] | 19 [3.9 to 34.1] | 63 [43.0 to 83.0]

3. Secondary Outcome: Tumor Response to Radiation Therapy for Patients With Medulloblastoma
Description: Percentages of patients with responses after radiation therapy (induction therapy) are reported with 95% confidence intervals. Complete and partial responses were considered responses.
Time Frame: 12 weeks after treatment initiation
Population: 83 of 87 eligible Arm A medulloblastoma patients were evaluated for response after induction, as were 85/89, 48/53, and 55/56 arm B, C, and D patients, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients)
Number analyzed (Participants) | 83 | 85 | 48 | 55
percentage of patients | 75.9 [65.3 to 84.6] | 78.8 [68.6 to 86.9] | 72.9 [58.2 to 84.7] | 81.8 [69.1 to 90.9]

4. Secondary Outcome: Tumor Response to Radiation Therapy for Patients With Supratentorial Primitive Neuroectodermal Tumor (SPNET)
Description: Percentages of patients with responses after radiation therapy (induction therapy) are reported with 95% confidence intervals. Complete and partial responses were considered responses. SPNET is no longer recognized by WHO (World Health Organization) as a disease entity. Additional trial information can be found under PubMed® # 30332335.
Time Frame: 12 weeks after treatment initiation
Population: 23 of 23 eligible Arm A SPNET patients were evaluated for response after induction, as were 18/19, 21/21, and 19/22 arm B, C, and D patients, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 23 | 18 | 21 | 19
percentage of patients | 69.9 [47.1 to 86.8] | 83.3 [58.6 to 96.4] | 66.7 [43.0 to 85.4] | 73.7 [48.8 to 90.9]

5. Secondary Outcome: Percent Probability of Overall Survival (OS) for Patients With Medulloblastoma
Description: The Kaplan-Meier method will be used to estimate 5-year OS, defined as the time from study enrollment to death from any cause, or to date of last contact. Estimates are reported with 95% confidence intervals. Data below represents all molecular subgroups combined.
Time Frame: Up to 5 years
Population: Eligible medulloblastoma patients are included.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients)
Number analyzed (Participants) | 87 | 89 | 53 | 56
Percent Probability | 66.0 [52.7 to 79.3] | 75.9 [64.1 to 87.7] | 69.9 [57.1 to 82.1] | 81.6 [70.8 to 92.4]

6. Secondary Outcome: Percent Probability of Overall Survival (OS) for Patients With Supratentorial Primitive Neuroectodermal Tumor (SPNET)
Description: The Kaplan-Meier method will be used to estimate 5-year OS, defined as the time from study enrollment to death from any cause, or to date of last contact.
Time Frame: Up to 5 years
Population: Eligible SPNET patients are included.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 23 | 19 | 21 | 22
Percent Probability | 60.9 [41.7 to 80.1] | 57.9 [35.8 to 80.0] | 35.3 [15.7 to 54.9] | 77.0 [59.4 to 94.6]

7. Secondary Outcome: The Estimated Full-scale IQ (FSIQ) at 9+/-3 Months Post Diagnosis for Medulloblastoma Patients
Description: Post-treatment neurocognitive function was assessed. Full-scale IQ (FSIQ) is a representative measurement for neurocognitive function. FSIQ was measured by IQ tests. Assessments within the time window, from eligible and evaluable patients are reported. The time window is 9+/-3 months post diagnosis, only the assessments before progression date were reported. The Range of FSIQ is 50-150. A higher FSIQ is better. Mean and standard deviation of FSIQ were calculated and reported.
Time Frame: 6 - 12 months post diagnosis
Population: Eligible medulloblastoma patients are included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients)
Number analyzed (Participants) | 22 | 30 | 13 | 23
Score on a scale | 96.6 (20.54) | 89.1 (17.45) | 83.5 (15.22) | 94.8 (16.88)

8. Secondary Outcome: The Estimated Full-scale IQ (FSIQ) at 30+/-6 Months Post Diagnosis for Medulloblastoma Patients
Description: Post-treatment neurocognitive function was assessed. Full-scale IQ (FSIQ) is a representative measurement for neurocognitive function. FSIQ was measured by IQ tests. Assessments within the time window, from eligible and evaluable patients are reported. The time window is 30+/-6 months post diagnosis, only the assessments before progression date were reported. The Range of FSIQ is 50-150. A higher FSIQ is better. Mean and standard deviation of FSIQ were calculated and reported.
Time Frame: 24 - 36 months post diagnosis
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: The Estimated Full-scale IQ (FSIQ) at 60+/-12 Months Post Diagnosis for Medulloblastoma Patients
Description: Post-treatment neurocognitive function was assessed. Full-scale IQ (FSIQ) is a representative measurement for neurocognitive function. FSIQ was measured by IQ tests. Assessments within the time window, from eligible and evaluable patients are reported. The time window is 60+/-12 months post diagnosis, only the assessments before progression date were reported. The Range of FSIQ is 50-150. A higher FSIQ is better. Mean and standard deviation of FSIQ were calculated and reported.
Time Frame: 48 - 72 months post diagnosis
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: The Estimated Full-scale IQ (FSIQ) at 9+/-3 Months Post Diagnosis for SPNET Patients
Description: as for outcome 7
Time Frame: 6 - 12 months post diagnosis
Population: Eligible SPNET patients are included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 7 | 4 | 9 | 7
Score on a scale | 84.6 (9.66) | 80.3 (28.86) | 99.3 (16.33) | 90.6 (21.9)

11. Secondary Outcome: The Estimated Full-scale IQ (FSIQ) at 30+/-6 Months Post Diagnosis for SPNET Patients
Description: as for outcome 8
Time Frame: 24 - 36 months post diagnosis
Population: Eligible SPNET patients are included
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 4 | 2 | 3 | 6
Score on a scale | 83.3 (9.98) | 57.5 (2.12) | 83.7 (4.04) | 88.5 (20.95)

12. Secondary Outcome: The Estimated Full-scale IQ (FSIQ) at 60+/-12 Months Post Diagnosis for SPNET Patients
Description: as for outcome 9
Time Frame: 48 - 72 months post diagnosis
Population: Eligible SPNET patients are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 5 | 1 | 2 | 3
score on a scale | 94.8 (15.55) | 48.0 (NA) — There is only one data available | 87.0 (5.66) | 79.7 (25.01)

13. Secondary Outcome: Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) at 9+/-3 Months Post Diagnosis for Medulloblastoma Patients
Description: Metacognition index (MI) was measured by BRIEF test. Assessments within the time window, from eligible and evaluable patients are reported. If the patient had disease progression, only the assessments before progression date were reported. The MI is a standard T- score, and it ranges from 0 to 100. The higher score reported suggests a higher level of dysfunction. Mean and standard deviation of MI were calculated and reported.
Time Frame: 6 - 12 months post diagnosis
Population: Eligible medulloblastoma patients are included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients)
Number analyzed (Participants) | 20 | 27 | 11 | 17
T-Score | 50.9 (11.32) | 50.2 (11.92) | 50.8 (10.04) | 47.5 (8.25)

14. Secondary Outcome: Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) at 30+/-6 Months Post Diagnosis for Medulloblastoma Patients
Description: Metacognition index (MI) was measured by BRIEF test. Assessments within the time window, from eligible and evaluable patients are reported. If the patient had disease progression, only the assessments before progression date were reported. The MI is a standard T- score, and it ranges from 0 to 100. The higher score reported suggests a higher level of dysfunction. Mean and standard deviation of MI were calculated and reported. SPNET is no longer recognized by WHO (World Health Organization) as a disease entity. Additional trial information can be found under PubMed® # 30332335.
Time Frame: 24 - 36 months post diagnosis
Reporting Status: Not Posted, anticipated posting 2025-12

15. Secondary Outcome: Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) at 60+/-12 Months Post Diagnosis for Medulloblastoma Patients
Description: as for outcome 13
Time Frame: 48 - 72 months post diagnosis
Reporting Status: Not Posted, anticipated posting 2025-12

16. Secondary Outcome: Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) at 9+/-3 Months Post Diagnosis for SPNET Patients
Description: as for outcome 13
Time Frame: 6 - 12 months post diagnosis
Population: Eligible SPNET patients are included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 4 | 3 | 7 | 4
T-Score | 53.8 (15.73) | 66.7 (1.53) | 46.1 (8.28) | 64.3 (6.5)

17. Secondary Outcome: Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) at 30+/-6 Months Post Diagnosis for SPNET Patients
Description: as for outcome 13
Time Frame: 24 - 36 months post diagnosis
Population: Eligible SPNET patients are included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 4 | 2 | 2 | 4
T-Score | 53.5 (8.27) | 75.5 (12.02) | 64.5 (2.12) | 53.5 (7.55)

18. Secondary Outcome: Metacognition Index (MI) on the Behavior Rating Inventory of Executive Function (BRIEF) at 60+/-12 Months Post Diagnosis for SPNET Patients
Description: as for outcome 13
Time Frame: 48 - 72 months post diagnosis
Population: Eligible SPNET patients are included.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
Number analyzed (Participants) | 2 | 1 | 2 | 3
T-Score | 56.0 (0) | 64.0 (NA) — There is only one data available | 71.5 (10.61) | 53.7 (21.2)

ADVERSE EVENTS:
Time Frame: While patients were on protocol therapy (including induction, 6 cycles of maintenance and 6 cycles of continuation) or up to 10 years while in follow-up
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Regimen A (Medulloblastoma Patients) | Regimen B (Medulloblastoma Patients) | Regimen C (Medulloblastoma Patients) | Regimen D (Medulloblastoma Patients) | Regimen A (SPNET Patients) | Regimen B (SPNET Patients) | Regimen C (SPNET Patients) | Regimen D (SPNET Patients)
All-Cause Mortality (participants affected / at risk) | 24/87 | 23/89 | 22/53 | 16/56 | 11/23 | 8/19 | 14/21 | 8/22
Serious Adverse Events (participants affected / at risk) | 7/87 | 11/89 | 5/53 | 6/56 | 2/23 | 0/19 | 1/21 | 0/22
Other Adverse Events (participants affected / at risk) | 72/87 | 80/89 | 47/53 | 52/56 | 21/23 | 18/19 | 18/21 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Medulloblastoma Patients) (N=87) | Regimen B (Medulloblastoma Patients) (N=89) | Regimen C (Medulloblastoma Patients) (N=53) | Regimen D (Medulloblastoma Patients) (N=56) | Regimen A (SPNET Patients) (N=23) | Regimen B (SPNET Patients) (N=19) | Regimen C (SPNET Patients) (N=21) | Regimen D (SPNET Patients) (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Medulloblastoma Patients) (N=87) | Regimen B (Medulloblastoma Patients) (N=89) | Regimen C (Medulloblastoma Patients) (N=53) | Regimen D (Medulloblastoma Patients) (N=56) | Regimen A (SPNET Patients) (N=23) | Regimen B (SPNET Patients) (N=19) | Regimen C (SPNET Patients) (N=21) | Regimen D (SPNET Patients) (N=22)
Neutrophil count decreased (Investigations) | 52 (113) | 59 (143) | 38 (82) | 40 (99) | 14 (31) | 16 (43) | 11 (21) | 16 (35)
White blood cell decreased (Investigations) | 49 (116) | 53 (124) | 37 (76) | 36 (88) | 12 (24) | 14 (35) | 12 (25) | 11 (26)
Platelet count decreased (Investigations) | 45 (88) | 65 (133) | 32 (63) | 42 (82) | 14 (21) | 17 (44) | 11 (16) | 14 (31)
Anemia (Blood and lymphatic system disorders) | 43 (81) | 59 (106) | 26 (52) | 32 (60) | 16 (25) | 14 (35) | 10 (16) | 15 (25)
Lymphocyte count decreased (Investigations) | 31 (79) | 32 (81) | 21 (44) | 15 (46) | 9 (21) | 10 (25) | 8 (18) | 7 (22)
Hypokalemia (Metabolism and nutrition disorders) | 23 (33) | 29 (41) | 17 (27) | 16 (25) | 5 (5) | 9 (11) | 4 (4) | 9 (11)
Febrile neutropenia (Blood and lymphatic system disorders) | 22 (38) | 45 (80) | 17 (25) | 21 (31) | 9 (9) | 13 (22) | 4 (4) | 8 (14)
Anorexia (Metabolism and nutrition disorders) | 19 (30) | 31 (46) | 12 (18) | 15 (24) | 3 (5) | 8 (14) | 6 (10) | 10 (13)
Nausea (Gastrointestinal disorders) | 13 (19) | 10 (12) | 9 (14) | 14 (18) | 3 (3) | 6 (11) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (18) | 10 (11) | 14 (18) | 8 (10) | 2 (2) | 6 (11) | 3 (3) | 5 (6)
Hearing impaired (Ear and labyrinth disorders) | 12 (13) | 11 (11) | 7 (16) | 6 (8) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 11 (27) | 27 (45) | 11 (19) | 14 (18) | 9 (10) | 7 (9) | 5 (5) | 8 (14)
Weight loss (Investigations) | 10 (12) | 9 (11) | 8 (9) | 5 (5) | 6 (9) | 3 (3) | 6 (9) | 4 (5)
Peripheral motor neuropathy (Nervous system disorders) | 8 (10) | 15 (20) | 6 (9) | 6 (8) | 1 (1) | 1 (1) | 3 (4) | 4 (8)
Hyponatremia (Metabolism and nutrition disorders) | 7 (8) | 8 (8) | 3 (4) | 2 (2) | 2 (2) | 2 (3) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 7 (7) | 6 (6) | 3 (5) | 2 (2) | 5 (8) | 4 (4) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (7) | 9 (10) | 3 (4) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 5 (5) | 3 (3) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4) | 3 (5) | 4 (5) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 4 (6)
Catheter related infection (Infections and infestations) | 4 (4) | 4 (4) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 4 (4) | 7 (9) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (7) | 3 (4) | 2 (2) | 1 (1) | 4 (6) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (2)
Skin infection (Infections and infestations) | 3 (3) | 5 (7) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 1 (2) | 1 (1) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 7 (8) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Ataxia (Nervous system disorders) | 2 (2) | 4 (6) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 2 (3) | 4 (5) | 2 (3) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (6) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (2) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mobitz type I (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cranial nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Azoospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalomyelitis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IVth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT00392327/Prot_SAP_000.pdf